CLINICAL TRIAL: NCT05503693
Title: A Single-center Randomized Double-blind Placebo-controlled Study to Investigate the Safety Tolerability and PK of SAD and MAD of AP303 Following Oral Administration and the Effect of Food on the PK of AP303 in Healthy Subjects
Brief Title: A Safety, Tolerability, and Pharmacokinetics Study of AP303 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alebund Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Alebund Pharmaceuticals (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP303-PK-01
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Healthy Subjects
Keywords: Safety, Tolerability, Pharmacokinetics, AP303, Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP303 (Experimental): AP303
  Interventions: Drug: AP303 50 μg; Drug: AP303 150 μg; Drug: AP303 300 μg; Drug: AP303 600 μg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo 50 μg; Drug: Placebo 150 μg; Drug: Placebo 300 μg; Drug: Placebo 600 μg

INTERVENTIONS:
Drug: AP303 50 μg — AP303 tablet
  Arms: AP303
Drug: AP303 150 μg — AP303 tablet
  Arms: AP303
Drug: AP303 300 μg — AP303 tablet
  Arms: AP303
Drug: AP303 600 μg — AP303 tablet
  Arms: AP303
Drug: Placebo 50 μg — Placebo tablet
  Arms: Placebo
Drug: Placebo 150 μg — Placebo tablet
  Arms: Placebo
Drug: Placebo 300 μg — Placebo tablet
  Arms: Placebo
Drug: Placebo 600 μg — Placebo tablet
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, first-in-human study in which the safety, tolerability, and pharmacokinetics of orally administered AP303 will be assessed in healthy adult subjects.

DETAILED DESCRIPTION:
The study will consist of 2 parts: Part A is a single ascending doses (SAD) phase enrolling a total of 4 cohorts of healthy subjects; Part B is a multiple ascending doses (MAD) phase enrolling 3 cohorts of healthy subjects. One cohort of Part A will receive AP303 under both fasted and fed conditions to investigate the effect of food.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, 18 to 55 years of age, inclusive.
2. Body Mas index(BMI) between 18 to 32 kg/m2 inclusive.
3. Female subjects of child-bearing potential must have a negative pregnancy test result and agree to use highly effective contraception consisting of two forms of birth control
4. Subjects and their partners of childbearing potential must use two medically approved methods of contraception and the subjects should refrain from sperm/egg donation for the duration of the study and for 3 months after drug administration

Exclusion Criteria:

1. Pregnant (positive pregnancy test) or lactating women, and male subjects with partners who are or plan to be pregnant or lactating.
2. History or symptoms of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, ophthalmologic, hematological or allergic disease, metabolic disorder, cancer or cirrhosis.
3. People with a history of specific allergies, or allergic conditions or known allergies to any ingredient of the investigational medicinal product (IMP).
4. History of having received or currently receiving any systemic anti-neoplastic or immune-modulatory treatment ≤ 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
5. Positive test at screening of any of the following: Hepatitis B (HBsAg), Hepatitis C (HCVAb) or human immunodeficiency virus (HIV Ab).
6. Received an investigational drug within 30 days or 5 xT1/2 whichever is longer prior to the first dose of our study for small molecule; or within 90 days or 5 x T1/2 whichever is longer prior to the first dose of our study drug; or device study within 90 days prior to screening or more than 4 times per year.
7. History of drug and/or alcohol abuse or addiction.
8. Use of >5 cigarettes or equivalent nicotine-containing product per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Single Dose and Food Effect Safety Outcome Measures | From baseline to Day 14 (Day 29 for Food Effect)
  Incidence and severity of adverse events (AEs), laboratory, ECG, and vital sign changes
Multiple Dose Safety Outcome Measures | From baseline to Day 28
  Incidence and severity of AEs, laboratory, ECG, and vital sign changes.
Cmax after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
Tmax after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
AUC0-last after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
AUC0-inf after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
t1/2 after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
CL/F after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
Ae and CLR (if warranted) after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
V/F after single dose | Pre-dose to 96 hours post-dose
  PK characteristics after single dose
Cmax after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
Tmax after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
AUC0-τ after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
Cav after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
t1/2 after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
Rac after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
Ae and CLR (if warranted) after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
V/F after multiple dose | Pre-dose to 12 hours post dose on Day 1; pre-dose to 96 hours post-dose on Day 14
  PK characteristics after multiple dose
Ctrough after multiple dose | Pre-dose on Days 2, 3, 4, 5, 7, 12, and 13
  PK characteristics after multiple dose

SECONDARY OUTCOMES:
Effect of Food on the single dose Cmax | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose Tmax | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose AUC0-last | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose AUC0-inf | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose t1/2 | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose CL/F | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose Ae and CLR (if warranted) | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK
Effect of Food on the single dose V/F | Pre-dose to 96 hours post-dose
  Effect of food on the single dose PK

CONTACTS AND LOCATIONS:
Overall Officials: Sam Francis, Doctor, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia